CLINICAL TRIAL: NCT06453928
Title: Starting Technology in At Risk Type 1 Diabetes (STAR-T1D) Study
Brief Title: Starting Technology in At Risk Type 1 Diabetes Study
Acronym: STAR-T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Principal Investigator, Estelle M. Everett, MD, MHS, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-000236; 5K23DK132482-02 (NIH)
Record Dates: First submitted 2024-04-26; First posted 2024-06-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Glucose Monitoring; Insulin Pump; Hybrid Closed Loop Systems; Diabetes Technology; Health Disparities
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hybrid Closed Loop Insulin Pump System (Experimental): Participants will meet 1:1 with our CDE for at least 6 sessions over 6 weeks. Sessions will cover self-management basics, carb counting, CGM interpretation, hypoglycemia and hyperglycemia management and troubleshooting device issues. The investigators will follow up with participants in 24 and 72 hours after CGM and insulin pump initiation, respectively, to answer any device related questions that may arise in between sessions.
  Participants will follow up at intervals of 1-4 weeks throughout the study. During visits, the investigators will assess for adherence and adverse effects and evaluate device and safety issues associated with pump settings in the HCL arm. The investigators will repeat A1c at 12 weeks and 24 weeks and administer follow up questionnaires at 12 and 24 weeks.
  Interventions: Device: Hybrid Closed Loop Insulin Pump System
- Control (No Intervention): Participants in the control arm will receive diabetes education at a similar frequency as the intervention group. Diabetes education for the control group will be a combination of in-person visits with the CDE and telephone brief diabetes education sessions.
  Participants will follow up at intervals of 1-4 weeks throughout the study. During visits, the investigators will assess for adherence and adverse effects. The investigators will repeat A1c at 12 weeks and 24 weeks and administer follow up questionnaires at 12 and 24 weeks.

INTERVENTIONS:
Device: Hybrid Closed Loop Insulin Pump System — Patients will be started on an automated insulin delivery system.
  Arms: Hybrid Closed Loop Insulin Pump System

SUMMARY:
Diabetes technology has revolutionized T1D management, disparities in technology access are evident among racial-ethnic minorities, patients with lower socioeconomic status and those with poorly controlled T1D (A1c>8.5%). In order to examine whether diabetes technology can reduce diabetes care burdens and enhance outcomes among some of highest need patients, diabetes technology clinical trials must be expanded beyond the very select populations included in studies thus far (ie., mostly White, higher SES). Therefore, the investigators propose to perform a pilot RCT of hybrid closed-loop insulin pump therapy (HCL) in 40 diverse adult patients with poorly controlled T1D (HbA1c >8.5%) from the largest academic and safety net health systems in the Los Angeles region to determine the feasibility of a RCT in this population and identify facilitators and barriers of effective use of closed loop insulin pump therapy in patients with poorly controlled T1D.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* A1c >8.5%
* Not insulin pump user
* Primary language of English or Spanish
* Have medical insurance coverage

Exclusion Criteria:

* No measured A1c in the past year
* Have comorbidities that can result in inaccurate hemoglobin A1c
* Have cognitive, physical or mental impairment precluding diabetes technology use
* Limited life expectancy (<1 year)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of screened participants that are eligible | 6 months
  Eligible among screened, enrolled among eligible, excluded among screened (and why) based on screening, recruitment and enrollment data.
Proportion of enrolled participants that are randomized | 6 months
  Randomized among enrolled, and receiving allocated intervention among randomized.
Proportion of average time delay to enrollment | 6 months
  Average time delay from screening to enrollment.
Proportion of retention among participants randomized to the Intervention Group | 6 months
  Retention among participants receiving allocated intervention after being randomized and discontinued intervention among randomized.
Proportion of retention among participants randomized | 6 months
  Participants lost to follow-up among those initially randomized.
Proportion of retention among participants randomized | 6 months
  Retention rates by participants completing all research assessments among randomized.
Number of participants who adhere to assigned treatment | 6 months
  Treatment-specific adherence, Adherence to study protocol and Proportion of planned assessments that are completed.
  Fidelity, which pertains to guaranteeing that the intervention is delivered in accordance with the established protocol, will be summarized by study arms, and differences between arms will be examined using t-tests or two-sample tests of proportions as appropriate.
  Adherence, which relates to the extent to which participants follow the treatment and study protocol, as well as the proportion of planned assessments completed, will be summarized by study arms, and differences between arms will be examined using t-tests or two-sample tests of proportions as appropriate.

SECONDARY OUTCOMES:
Change in A1c | 6 months
  Serum Hemoglobin A1c laboratory measurement
Episodes and % of time with severe hypoglycemia ( BG <54 mg/dl) | 6 months
  Hypoglycemia will be measure by combining CGM metrics and glucometer to report severe hypoglycemia in mg/dl.
Mean Diabetes Ketoacidosis Episodes Incidence | 6 months
  Assess instances of diabetic ketoacidosis through participant surveys and comprehensive chart reviews.
ED visits/Hospitalizations Number of diabetes related ED visits or hospitalizations | 6 months
  Number of diabetes related ED visits or hospitalizations
Treatment Burden and Satisfaction: Diabetes Distress | 6 months
  Assessing treatment burden through the Type 1 Diabetes Distress Assessment System T1DDAS, which comprises eight questions and evaluates ten prevalent sources of diabetes distress in adults with type 1 diabetes. The score indicates the level of diabetes distress reported by the respondent, with higher scores indicating greater intensity. The core scale scoring ranges 1 to 5. This scale assesses each of ten common Sources of diabetes distress for adults with type 1 diabetes: Financial Worries, Interpersonal Challenges, Management Difficulties, Shame, Hypoglycemia Concerns, Healthcare Quality, Lack Of Diabetes Resources, Technology Challenges, Burden To Others, Worries About Complications. The higher the score, the more impactful that Source is likely to be in contributing to diabetes distress for this individual with the minimum value being 1 and maximum value being 5.
Treatment Burden and Satisfaction: Insulin Treatment Satisfaction | 6 months
  Assessed treatment burden and satisfaction using the Insulin Treatment Satisfaction Questionnaire (ITSQ), consisting of 22 questions among 5 content clusters with a score from 0 to 100% where a higher score indicates greater satisfaction with insulin treatment. The scale explores perceptions of current insulin treatment and its impact on daily life.
Treatment Burden and Satisfaction: Glucose Monitoring System Satisfaction (GMSS) | 6 months
  Examined treatment burden and satisfaction employing the Glucose Monitoring System Satisfaction Survey (GMSS), comprising 15 questions divided into four subcategories: openness, emotional burden, behavioral burden and trust. Higher scores within each subcategory denote either greater satisfaction or burden, depending on the specific aspect assessed with the minimum value being 1 and maximum value being 5. The total scare has a minimum value of 1 and maximum value of 15 with higher scores indicating greater satisfaction. The scores are obtained by calculating the mean for each.
Treatment Burden and Satisfaction: Motivation and Attitudes Towards Changing Health (MATCH) | 6 months
  Assessed treatment burden and satisfaction using the Motivation and Attitudes towards Health Scale (MATCH), consisting of nine questions categorized into four subgroups: willingness to make changes, perceived ability to make or maintain changes, feeling changes are worthwhile, and overall mean/average of willingness, able, and worthwhile. Scores are calculated by determining the mean or average response within each category with higher scores meaning a better outcome.
  WILLINGNESS: minimum value is 1 and maximum value is 5. ABLE: minimum value is 1 and maximum value is 5. WORTHWHILE: minimum value is 1 and maximum value is 5. TOTAL SCALE: minimum value is 1 and maximum value is 9.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCLA, Santa Monica, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Harbor-UCLA Medical Center, Torrance, California

IPD SHARING:
Plan to Share IPD: No